CLINICAL TRIAL: NCT05313373
Title: The Effect of Virtual Reality On Women's Perceptıons of Fear, Pain, Anxiety and Satisfaction Undergoing Hysterosalpingography; A Randomized Controlled Research
Brief Title: The Effect of Virtual Reality on Women Undergoing Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NESLİHAN YILMAZ SEZER (Other)
Responsible Party: Sponsor-Investigator, NESLİHAN YILMAZ SEZER, Faculty of Nursing, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 04/49
Record Dates: First submitted 2022-03-14; First posted 2022-04-06 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Hysterosalpingography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental)
  Interventions: Other: Virtual Reality
- Control Group (No Intervention)

INTERVENTIONS:
Other: Virtual Reality — In addition to the routine procedure, virtual reality glasses will be applied to the women in the virtual reality group of the research. Virtual reality glasses is a device that works on compatible smart mobile phones. After being taken to the gynecological table for the HSG procedure, the women included in the experimental group will be made to watch a video lasting an average of 10 minutes with virtual reality glasses until the procedure is completed. While watching the video, the relaxing music of the video will be played.
  Arms: Virtual Reality Group

SUMMARY:
The aim of this study is to determine the effect of virtual reality on perceived pain, anxiety, fear, physiological reactions and satisfaction in women during the HSG procedure.

Hypotheses H01; In the HSG procedure, there was no difference between the pain score of the virtual reality group and the pain score of the control group.

H02; In the HSG procedure, there was no difference between the anxiety score of the virtual reality group and the anxiety score of the control group.

H03; In the HSG procedure, there was no difference between the satisfaction score of the virtual reality group and the satisfaction score of the control group.

H04; In the HSG procedure, there was no difference between the vital signs of the virtual reality group and the control group.

H05; In the HSG procedure, there was no difference between the fear score of the virtual reality group and the fear score of the control group.

The study will be carried out in two different groups. The practice will start with meeting the women who apply to the Radiology clinic for an HSG. After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Virtual Reality Group In addition to the routine procedure, virtual reality glasses will be applied to the women in the virtual reality group of the research. Virtual reality glasses is a device that works on compatible smart mobile phones. After being taken to the gynecological table for the HSG procedure, the women included in the experimental group will be made to watch a video lasting an average of 10 minutes with virtual reality glasses until the procedure is completed. While watching the video, the relaxing music of the video will be played in the practice room with a bluetooth speaker.

Control Group Patients in the control group of the study will not be subjected to any treatment other than the routine procedure.

ELIGIBILITY:
Inclusion Criteria:

* primary infertility
* Agreeing to participate in the research and obtaining written permission,
* No hearing or vision problems
* The first time HSG procedure will be applied

Exclusion Criteria:

* Didn't watch the whole video
* Those with motion-sensitive diseases such as vertigo, meniere
* Using any pharmacological pain-reducing method within 30 minutes
* Difficulty in the HSG process or completing the process with more than one attempt
* Use of antidepressants or sedatives
* Any history of allergy to radio-opaque dye

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | immediately before the HSG procedure and immediately after the HSG procedure
  STAI-S consist of 20 items with four points Likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
Change in the degree of pain experienced during the procedure | immediately before the HSG procedure, and immediately after the HSG procedure, and 15 minutes after the HSG procedure
  The pain was assessed using 0-100 mm VAS for determining perceptions of pain during the procedure. This scale is widely used and has demonstrated reliability and validity in the measurement of acute pain. A high score on the scale indicated a high level of pain and a score of 0 pointed to no pain at all (Bijur, Silver, & Gallagher, 2001). Each participant was asked to mark her current level of perceived pain along the scale, with the number corresponding to the marked point recorded as the pain score
Change in fear | immediately before the HSG procedure, immediately after the HSG procedure, and 15 minutes after the HSG procedure
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "no fear at all" and the right end reads "the most intense fear possible". A high score on the scale indicated a high level of fear and a score of 0 pointed to no fear.

SECONDARY OUTCOMES:
the degree of satisfaction | 15 minutes after the HSG procedure
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "I am not satisfied at all" and the right end reads "very satisfied". A high score on the scale indicated a high level of satisfied and a score of 0 pointed to no satisfied.
Change in blood pressure | immediately before the HSG procedure, and immediately after the HSG procedure, and 15 minutes after the HSG procedure
  mmHg
Change in heart rate | immediately before the HSG procedure, and immediately after the HSG procedure, and 15 minutes after the HSG procedure
  beats per minute (bpm)
Change in body temperature | immediately before the HSG procedure, and immediately after the HSG procedure, and 15 minutes after the HSG procedure
  degrees Celsius
Change in the saturation of peripheral oxygen SpO2 | immediately before the HSG procedure, and immediately after the HSG procedure, and 15 minutes after the HSG procedure
HSG result | 15 minutes after the HSG procedure
  both tubes patent, one fallopian tubes occluded, both fallopian tubes occluded
contrast medium volume | during HSG prosedure
  milliliter (ml)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University Fertility Diagnosis, Treatment, Research and Application Center, Ankara, Mamak
  - Ankara University Fertility Diagnosis, Treatment, Research and Application Center, Ankara

IPD SHARING:
Plan to Share IPD: Undecided